CLINICAL TRIAL: NCT01970540
Title: Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of PM01183 in Combination With Doxorubicin in Non-heavily Pretreated Patients With Selected Advanced Solid Tumors
Brief Title: Study Escalating Doses of PM01183 in Combination With Fixed Doxorubicin in Patients With Specific Advanced Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-A-003-10
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-01

CONDITIONS: Endometrial Adenocarcinomas; Neuroendocrine Tumors; Small-cell Lung Cancer With Less Than 2 Prior Cytotoxic-containing Lines of Therapy
Keywords: lurbinectedin; PM01183; tumors; cancer; Pharma Mar
MeSH Terms: conditions — Neuroendocrine Tumors; Neoplasms | interventions — PM 01183; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lurbinectedin (PM01183) / doxorubicin (Experimental)
  Interventions: Drug: lurbinectedin (PM01183); Drug: Doxorubicin

INTERVENTIONS:
Drug: lurbinectedin (PM01183) — lurbinectedin (PM01183) is presented as powder for concentrate for solution for infusion with two strengths, 1-mg and 4-mg vials.
Drug: Doxorubicin — Commercially available presentations of vials containing doxorubicin will be provided as appropriate.

SUMMARY:
Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of PM01183 in Combination with Fixed Doxorubicin in Non- Heavily Pretreated Patients with Selected Advanced Solid Tumors to determine the maximum tolerated dose (MTD) and the recommended dose (RD) of PM01183 in combination with doxorubicin, to characterize the safety profile and feasibility of this combination, to characterize the pharmacokinetics (PK) of this combination, to obtain preliminary information on the clinical antitumor activity,to explore the feasibility, safety and efficacy of a potential improvable dose of this combination in selected tumor types [i.e. small cell lung cancer (SCLC) and endometrial cáncer] and to evaluate the pharmacogenomics (PGx) in tumor samples of patients exposed to PM01183 and doxorubicin at the RD in order to assess potential markers of response and/or resistance.

DETAILED DESCRIPTION:
The study has currently met its primary end point and is now recruiting patients to be treated at the RD expansion cohort of selected tumor types, specifically: endometrial adenocarcinomas, neuroendocrine tumors, and small-cell lung cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily written informed consent
* Age: between 18 and 75 years (both inclusive).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1. Cohort of patients with SCLC and endometrial cáncer ECOG PS ≤ 2.
* Life expectancy ≥ 3 months.
* Patients with a histologically/cytologically confirmed diagnosis of advanced disease of any of the following tumors:

  1. Breast cancer
  2. Soft-tissue sarcoma
  3. Primary bone sarcomas.
  4. Gynecologic tumors (endometrial adenocarcinomas, epithelial ovarian cancer...)
  5. Hepatocellular carcinoma
  6. Gastroenteropancreatic neuroendocrine tumors
  7. Small cell lung cancer (SCLC)
  8. Gastric cancer
  9. Bladder cancer
  10. Adenocarcinoma of unknown primary site
* At least three weeks since the last anticancer therapy, including radiotherapy
* Adequate bone marrow, renal, hepatic, and metabolic function
* Left ventricular ejection fraction (LVEF) by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan within normal range (according to institutional standards).
* Women of childbearing potential must have a negative serum pregnancy test before study entry. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for six weeks after discontinuation of treatment

Exclusion Criteria:

* Concomitant diseases/conditions:

  * History or presence of unstable angina, myocardial infarction, congestive heart failure, or clinically significant valvular heart disease within last year.
  * Symptomatic or any uncontrolled arrhythmia
  * Ongoing chronic alcohol consumption, or cirrhosis
  * Active uncontrolled infection.
  * Known human immunodeficiency virus (HIV) infection.
  * Any other major illness that, in the Investigator's judgment
* Brain metastases or leptomeningeal disease involvement.
* Men or women of childbearing potential who are not using an effective method of contraception
* Patients who have had radiation therapy in more than 35% of the bone marrow. This criterion will not apply to cohort of patients with SCLC and endometrial cáncer.
* History of previous bone marrow and/or stem cell transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-05-25 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (6):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Centro Oncológico Md Anderson International España, Madrid
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Fundación Instituto Valenciano de Oncología, Valencia
- UCLH (University College London Hospitals), London, United Kingdom

REFERENCES:
- [Derived] Olmedo ME, Forster M, Moreno V, Lopez-Criado MP, Brana I, Flynn M, Doger B, de Miguel M, Lopez-Vilarino JA, Nunez R, Kahatt C, Cullell-Young M, Zeaiter A, Calvo E. Efficacy and safety of lurbinectedin and doxorubicin in relapsed small cell lung cancer. Results from an expansion cohort of a phase I study. Invest New Drugs. 2021 Oct;39(5):1275-1283. doi: 10.1007/s10637-020-01025-x. Epub 2021 Mar 11. PMID 33704620

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 122 patients were enrolled at 7 sites. 120 patients were treated with DOX/PM01183 combination: 73 Cohort A (DOX [mg/m2]+PM01183 [mg FD]) & 47 Cohort B (DOX [mg/m2]+PM01183 [mg/m2]).
  Patients participated between 25May2011-9Aug2017 (last followup). First dose of the first cycle was given on 13Jun2011 and last dose of the last cycle on 19Jul2017
Pre-assignment Details: Screening details:
  Age 18-75;CI signed;ECOG PS≤1;histologically/cytologically confirmed diagnosis of advanced disease;Life expectancy≥3 months;not previously treated with anthracycline-containing therapy for advanced disease;No more than two prior lines of cytotoxic-containing chemotherapy regimens;CPK≤2.5xULN;Albumin≥2.5 g/dL
Groups:
- Cohort A: DOX: 50 mg/m² q3wk immediately followed by PM01183. The dose escalation scheme was: 3.0, 3.5, 5.0, 6.0, 7.0 mg FD
  lurbinectedin (PM01183): lurbinectedin (PM01183) is presented as powder for concentrate for solution for infusion with two strengths, 1-mg and 4-mg vials.
  Doxorubicin: Commercially available presentations of vials containing doxorubicin will be provided as appropriate.
- Cohort B: SCLC 2nd Line: Patients with SCLC 2nd line received the following on Day 1 q3wk (three weeks = one treatment cycle), administered: DOX 40 mg/m2 immediately followed by PM01183: 2.0 mg/m2.
  lurbinectedin (PM01183): lurbinectedin (PM01183) is presented as powder for concentrate for solution for infusion with two strengths, 1-mg and 4-mg vials.
  Doxorubicin: Commercially available presentations of vials containing doxorubicin will be provided as appropriate.
  SCLC, small cell lung cancer
- Cohort B: Endometrial: Patients with endometrial cancer received the following on Day 1 q3wk (three weeks = one treatment cycle), administered: DOX 40 mg/m2 immediately followed by PM01183: 2.0 mg/m2.
  lurbinectedin (PM01183): lurbinectedin (PM01183) is presented as powder for concentrate for solution for infusion with two strengths, 1-mg and 4-mg vials.
  Doxorubicin: Commercially available presentations of vials containing doxorubicin will be provided as appropriate.
Period: Overall Study
Arm/Group | Cohort A | Cohort B: SCLC 2nd Line | Cohort B: Endometrial
Started | 73 | 28 | 19
Completed | 0 | 0 | 0
Not Completed | 73 | 28 | 19
Not completed — Non-treatment-related AE | 0 | 0 | 1
Not completed — Progressive disease | 55 | 23 | 10
Not completed — Treatment delay over protocol | 0 | 0 | 1
Not completed — Physician Decision | 7 | 2 | 0
Not completed — Clinical progression | 0 | 1 | 1
Not completed — End of study | 2 | 0 | 2
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Treatment-related AE | 4 | 0 | 2
Not completed — Withdrawal by Subject | 4 | 0 | 1
Not completed — Clinical deterioration | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort A: DOX: 50 mg/m² q3wk immediately followed by PM01183. The dose escalation scheme was: 3.0, 3.5, 5.0, 6.0, 7.0 mg FD
- Cohort B: SCLC 2nd Line: Patients with SCLC 2nd line received the following on Day 1 q3wk (three weeks = one treatment cycle), administered: DOX 40 mg/m2 Immediately followed by PM01183: 2.0 mg/m2.
- Cohort B: Endometrial: Patients with endometrial cancer received the following on Day 1 q3wk (three weeks = one treatment cycle), administered: DOX 40 mg/m2 immediately followed by PM01183: 2.0 mg/m2.
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B: SCLC 2nd Line | Cohort B: Endometrial | Total
Number analyzed (Participants) | 73 | 28 | 19 | 120
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 0 | 0 | 0 | 0
  Age: Between 18 and 65 years | 53 | 18 | 8 | 79
  Age: >=65 years | 20 | 10 | 11 | 41
Age, Continuous [Median (Full Range); unit: years] | 62.2 [22 to 78] | 64 [49 to 77] | 66 [55 to 73] | 62.2 [22 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 7 | 19 | 64
  Male | 35 | 21 | 0 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race : Caucasian | 72 | 27 | 19 | 118
  Race : Asian/oriental | 1 | 0 | 0 | 1
  Race : Black | 0 | 1 | 0 | 1
ECOG PS [Count of Participants; unit: Participants] — ECOG PS, Eastern Cooperative Oncology Group performance status PS 0 Fully active able to carry on all pre-disease performance without restriction PS 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature PS 2 Ambulatory and capable of all selfcare but unable to carry out any work activities up and about more than 50% of waking hours PS 3 Capable of only limited selfcare confined to bed or chair more than 50% of waking hours PS 4 Completely disabled cannot carry on any selfcare; totally confined to bed or chair PS 5 Dead
  Participants
    PS 0 | 27 | 9 | 6 | 42
    PS 1 | 46 | 19 | 12 | 77
    PS 2 | 0 | 0 | 1 | 1
Tumor type [Count of Participants; unit: Participants] — ET-GEP, neuroendocrine-gastroenteropancreatic tumor; SCLC, small cell lung cancer; STS, soft tissue sarcoma; HCC, hepatocellular carcinoma
  Participants
    SCLC 2 line | 22 | 28 | 0 | 50
    SCLC 3 line | 6 | 0 | 0 | 6
    Endometrial | 15 | 0 | 19 | 34
    NET-GEP | 8 | 0 | 0 | 8
    STS | 8 | 0 | 0 | 8
    Bladder | 5 | 0 | 0 | 5
    Gastric | 4 | 0 | 0 | 4
    Breast | 3 | 0 | 0 | 3
    Ovarian | 1 | 0 | 0 | 1
    HCC | 1 | 0 | 0 | 1
Lines of prior anticancer therapies [Count of Participants; unit: Participants]
  0 lines | 12 | 0 | 3 | 15
  1 line | 42 | 27 | 11 | 80
  2 lines | 16 | 1 | 5 | 22
  3 lines | 2 | 0 | 0 | 2
  >3 lines | 1 | 0 | 0 | 1
Body surface area [Median (Full Range); unit: m^2] | 1.8 [1.3 to 2.3] | 1.9 [1.5 to 2.3] | 1.8 [1.6 to 2.3] | 1.8 [1.3 to 2.3]
Time from diagnosis to first infusion [Median (Full Range); unit: months] | 16.2 [3.0 to 277.8] | 8.4 [3.9 to 19.8] | 22.0 [10.6 to 79.2] | 16.2 [3.0 to 277.8]
Time from last progressive disease to first infusion [Median (Full Range); unit: months] | 0.9 [0.1 to 3] | 0.9 [0.2 to 3.4] | 1.3 [0.6 to 4.2] | 0.9 [0.1 to 4.2]
Time to progression of last prior therapy [Median (Full Range); unit: months] | 6.3 [1.2 to 34.3] | 6.8 [1 to 18.9] | 7.1 [1.1 to 22.6] | 6.7 [1 to 34.3]
Sites of disease at baseline [Median (Full Range); unit: number of sites] | 2 [1 to 6] | 3 [1 to 6] | 2 [1 to 3] | 2 [1 to 6]
Lines of prior anticancer therapies [Median (Full Range); unit: lines of therapies] | 1 [0 to 4] | 1 [1 to 2] | 1 [0 to 2] | 1 [0 to 4]
Agents of prior anticancer therapies [Median (Full Range); unit: Agents therapies] | 2 [0 to 6] | 2 [2 to 3] | 2 [0 to 4] | 2 [0 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: A minimum of three patients will be included at each DL. If no patients experience a DLT during Cycle 1, the dose will be escalated. If one of three patients experiences a DLT, three additional patients will be included at that level. If >1 evaluable patient during dose escalation at a given DL experience a DLT during Cycle 1, that DL will be considered the MTD and dose escalation will be terminated, except if all DLTs are related to neutropenia exclusively, in which case dose escalation may be resumed as originally planned in a new cohort of patients but with compulsory primary G-CSF prophylaxis.
Time Frame: During the first cycle of treatment, up to 28 days
Population: Fifty-seven of the 61 patients treated in this cohort without primary G-CSF prophylaxis were evaluable for DLTs Eleven of the 12 patients treated with primary G-CSF prophylaxis in this cohort were evaluable for DLTs.
Measure: Number; unit: DOX mg/m2 PM01183 mg FD
Groups:
- Patients Without Primary G-CSF Prophylaxis: All participants who received at least one complete cycle study treatments without Primary G-CSF Prophylaxis
- Patients With Primary G-CSF Prophylaxis: All participants who received at least one complete cycle study treatments with Primary G-CSF Prophylaxis
Arm/Group | Patients Without Primary G-CSF Prophylaxis | Patients With Primary G-CSF Prophylaxis
Number analyzed (Participants) | 57 | 11
DOX mg/m2 PM01183 mg FD
  Doxorubicin | 50 | 50
  PM01183 | 5.0 | 5.0

2. Primary Outcome: Recommended Dose (RD)
Description: The DL immediately below the MTD, or DL4 if the MTD is not yet defined during dose escalation before the last DL (i.e., DL4) is reached, was to be initially expanded up to a minimum of nine evaluable patients. If less than three among the first nine evaluable patients treated within the expansion cohort experience a DLT during Cycle 1, this DL will be the RD.
Time Frame: During the first cycle of treatment, up to 28 days
Population: Fifty-seven of the 61 patients treated in this cohort without primary G-CSF prophylaxis were evaluable for DLTs
Measure: Number; unit: DOX mg/m2 PM01183 mg FD
Arm/Group | Patients Without Primary G-CSF Prophylaxis
Number analyzed (Participants) | 57
DOX mg/m2 PM01183 mg FD
  Doxorubicin | 50
  PM01183 | 4.0

3. Primary Outcome: Number of Participants With Dose-limiting Toxicities
Description: DLT,dose-limiting toxicity Patients enrolled into this study were originally not allowed to receive primary G-CSF prophylaxis. However, the finding of dose-limiting febrile neutropenia in two patients treated at dose level I in the present study (see below) suggested that increasing doses of the DOX/PM01183 combination might require primary G-CSF prophylaxis to decrease the risk of febrile neutropenia. Therefore, a separate dose escalation was established to define the MTD and the RD of the DOX/PM01183 combination with compulsory primary G-CSF prophylaxis.
Time Frame: During the first cycle of treatment, up to 28 days
Population: Patients evaluable for the primary endpoint (evaluable for DLT): 5 patients were not evaluable in Cohort A and 1 patient in Cohort B.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Dose I Without Primary G-CSF Prophylaxis: DOX 50 mg/m2 plus PM01183 3.5 mg FD without primary G-CSF prophylaxis
- Cohort A: Dose II Without Primary G-CSF Prophylaxis: DOX 50 mg/m2 plus PM01183 3.0 mg FD without primary G-CSF prophylaxis
- Cohort A: Dose I Without Primary G-CSF Proph and Age Limit: DOX 50 mg/m2 plus PM01183 3.5 mg FD and the Investigators and the Sponsor decided to amend the study's eligibility criteria, which originally did not establish a maximum age limit for the patients, in order to restrict accrual to patients aged between 18 and 75 years, both inclusive
- Cohort A: Dose III Without Primary G-CSF Prophylaxis: DOX 50 mg/m2 plus PM01183 4.0 mg FD without primary G-CSF prophylaxis
- Cohort A: Dose IV Without Primary G-CSF Prophylaxis: DOX 50 mg/m2 plus PM01183 5.0 mg FD without primary G-CSF prophylaxis
- Cohort A: Dose I With Primary G-CSF Prophylaxis: DOX 50 mg/m2 plus PM01183 3.5 mg FD. Patients enrolled into this study were originally not allowed to receive primary G-CSF prophylaxis.
  However, the finding of dose-limiting febrile neutropenia in two patients treated at dose level I (DOX 50 mg/m2 plus PM01183 3.5 mg FD) in the present study suggested that increasing doses of the DOX/PM01183 combination might require primary G-CSF prophylaxis to decrease the risk of febrile neutropenia. Therefore, a separate dose escalation was established to define the MTD and the RD of the DOX/PM01183 combination with compulsory primary G-CSF prophylaxis
- Cohort A: Dose III With Primary G-CSF Prophylaxis: DOX 50 mg/m2 plus PM01183 4.0 mg FD Patients enrolled into this study were originally not allowed to receive primary G-CSF prophylaxis.
  However, the finding of dose-limiting febrile neutropenia in two patients treated at dose level I (DOX 50 mg/m2 plus PM01183 3.5 mg FD) in the present study suggested that increasing doses of the DOX/PM01183 combination might require primary G-CSF prophylaxis to decrease the risk of febrile neutropenia. Therefore, a separate dose escalation was established to define the MTD and the RD of the DOX/PM01183 combination with compulsory primary G-CSF prophylaxis
- Cohort A: Dose IV With Primary G-CSF Prophylaxis: DOX 50 mg/m2 plus PM01183 5.0 mg FD Patients enrolled into this study were originally not allowed to receive primary G-CSF prophylaxis.
  However, the finding of dose-limiting febrile neutropenia in two patients treated at dose level I (DOX 50 mg/m2 plus PM01183 3.5 mg FD) in the present study suggested that increasing doses of the DOX/PM01183 combination might require primary G-CSF prophylaxis to decrease the risk of febrile neutropenia. Therefore, a separate dose escalation was established to define the MTD and the RD of the DOX/PM01183 combination with compulsory primary G-CSF prophylaxis
- Cohort B: DOX [mg/m2] Plus PM01183 [mg/m2]: DOX [mg/m2] plus PM01183 [mg/m2] Patient accrual into Cohort B started after the RD for the DOX/PM01183 combination had been defined in Cohort A. The dose evaluated in Cohort B was based on this RD, but the DOX dose was decreased to 40 mg/m2 and the PM01183 dose was changed to a BSA-based dose of 2.0 mg/m2 in order to improve the feasibility of this combination in patients with SCLC treated as second-line therapy and in patients with endometrial cancer. In accordance with the findings obtained in Cohort A, no patients in Cohort B received primary G-CSF prophylaxis.
Arm/Group | Cohort A: Dose I Without Primary G-CSF Prophylaxis | Cohort A: Dose II Without Primary G-CSF Prophylaxis | Cohort A: Dose I Without Primary G-CSF Proph and Age Limit | Cohort A: Dose III Without Primary G-CSF Prophylaxis | Cohort A: Dose IV Without Primary G-CSF Prophylaxis | Cohort A: Dose I With Primary G-CSF Prophylaxis | Cohort A: Dose III With Primary G-CSF Prophylaxis | Cohort A: Dose IV With Primary G-CSF Prophylaxis | Cohort B: DOX [mg/m2] Plus PM01183 [mg/m2]
Number analyzed (Participants) | 5 | 7 | 3 | 37 | 5 | 3 | 3 | 5 | 46
Participants | 2 | 0 | 0 | 8 | 2 | 0 | 0 | 2 | 4

4. Secondary Outcome: Best Overall Tumor Response
Description: Tumor response was evaluated according to the RECIST v.1.1 for target lesions and assessed by computed tomography (CT) scans or magnetic resonance imagings (MRIs): Progressive disease (PD) is declared when there is an increase in sum of target disease ≥ 20%, stable diease (SD) when the change is > -30% and ≤ 20%, partial response (PR) when there is a decrease in sum of target disease ≥ 30%, and complete response (CR) when all lesions have disappeared or all lesions have disapeared and all nodal disease is < 10 mm each.
Time Frame: Tumor assessments were done every six weeks up to study completion
Population: Cohort A: 1 patient of 73 was not evaluable: extensive bone marrow involvement
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B: SCLC 2nd Line: Patients with SCLC 2nd line received the following on Day 1 q3wk (three weeks = one treatment cycle), administered: DOX 40 mg/m2 immediately followed by PM01183: 2.0 mg/m2.
  lurbinectedin (PM01183): lurbinectedin (PM01183) is presented as powder for concentrate for solution for infusion with two strengths, 1-mg and 4-mg vials.
  Doxorubicin: Commercially available presentations of vials containing doxorubicin will be provided as appropriate.
Arm/Group | Cohort A | Cohort B: SCLC 2nd Line | Cohort B: Endometrial
Number analyzed (Participants) | 72 | 28 | 19
Participants
  CR | 7 | 1 | 0
  PR | 19 | 9 | 8
  SD≥4 months | 13 | 4 | 4
  SD<4 months | 11 | 6 | 3
  PD | 22 | 8 | 4

5. Secondary Outcome: Duration of Response
Description: The duration of overall response was measured from the time measurement criteria are met for complete response (CR)/ PR, whichever is first recorded, until the first date in which progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started) or the date of death. In absence of disease progression or death, the duration of response was censored on the date of last tumor evaluation.
Time Frame: Time from the time measurement criteria are met for complete response, whichever is first recorded, until the first date in which progressive disease is objectively documented or the date of death, assessed up to 72 months
Population: Cohort A: 26 patients showed response to treatment Events: 26 (100.0%) Cohort B SCLC: 10 patients showed response to treatment Events: 10 (100.0%) Cohort B: Endometrial: 8 patients showed response to treatment Events: 4 (50.0%)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B: SCLC 2nd Line | Cohort B: Endometrial
Number analyzed (Participants) | 26 | 10 | 8
months | 7.2 [3.4 to 8.6] | 5.2 [1 to 6.9] | 7.5 [6.4 to NA] — Not reached

6. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time from the date of first infusion of study treatment to the date of progression or death (due to any cause). If progression or death has not occurred at the time of the analysis, the PFS was censored on the date of last tumor evaluation.
Time Frame: Time from the date of first administration to the date of PD or death (of any cause), whichever came first, assessed up to 72 months
Population: Cohort A: 1 patient was not evaluable: extensive bone marrow involvement Events: 66 (91.7%) Cohort B: SCLC Events: 28 (100.0%) Cohort B: Endometrial: Events: 14 (73.7%)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B: SCLC 2nd Line | Cohort B: Endometrial
Number analyzed (Participants) | 72 | 28 | 19
months | 3.8 [2.6 to 5.3] | 3.3 [1.4 to 6.2] | 7.7 [2.0 to 16.7]

7. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from the date of first infusion of study treatment to the date of death (due to any cause). Patients with no documented death were censored at the last date they are known to be alive
Time Frame: Time from the date of first administration to the date of death (of any cause), assessed up to 72 months
Population: Cohort A: Events: 15 (20.5%); Cohort B: SCLC: Events: 22 (78.6%); Cohort B: Endometrial Events: 11 (57.9%)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B: SCLC 2nd Line | Cohort B: Endometrial
Number analyzed (Participants) | 73 | 28 | 19
months | 36.9 [15.1 to NA] — Not reached | 7.9 [4.2 to 11.5] | 14.2 [4.5 to NA] — Not reached

ADVERSE EVENTS:
Time Frame: Participants were assessed through study completion, approximately 6 years
Description: All 120 patients treated in this study were evaluable for safety
Groups:
- Cohort A: 73 patients treated in Cohort A (DOX [mg/m2] plus PM01183 [mg FD]) were evaluable for safety
Arm/Group | Cohort A | Cohort B: SCLC 2nd Line | Cohort B: Endometrial
All-Cause Mortality (participants affected / at risk) | 15/73 | 22/28 | 11/19
Serious Adverse Events (participants affected / at risk) | 47/73 | 19/28 | 14/19
Other Adverse Events (participants affected / at risk) | 73/73 | 28/28 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=73) | Cohort B: SCLC 2nd Line (N=28) | Cohort B: Endometrial (N=19)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Acute monocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 25 (32) | 4 (4) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 9 (12) | 2 (5) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (10) | 4 (11) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Trigeminal nerve disorder (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Neutropenic infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=73) | Cohort B: SCLC 2nd Line (N=28) | Cohort B: Endometrial (N=19)
Hypotensions (Vascular disorders) | 6 (8) | 3 (3) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 33 (67) | 7 (15) | 1 (1)
Chest pain (General disorders) | 6 (9) | 1 (1) | 3 (3)
Chills (General disorders) | 4 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 66 (382) | 25 (118) | 17 (111)
Infusion site reaction (General disorders) | 4 (6) | 0 (0) | 1 (2)
Malaise (General disorders) | 4 (5) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 34 (110) | 5 (19) | 5 (12)
Oedema peripheral (General disorders) | 7 (13) | 1 (1) | 3 (7)
Pain (General disorders) | 4 (4) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 24 (35) | 5 (6) | 3 (3)
Anxiety (Psychiatric disorders) | 10 (15) | 3 (4) | 3 (7)
Confusional state (Psychiatric disorders) | 4 (5) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 13 (24) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 9 (9) | 3 (6) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 1 (1)
Weight decreased (Investigations) | 15 (26) | 6 (7) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (5) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (73) | 14 (19) | 6 (14)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 (52) | 11 (34) | 5 (10)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (13) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 39 (99) | 7 (26) | 5 (10)
Neutropenia (Blood and lymphatic system disorders) | 31 (75) | 10 (20) | 7 (60)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (14) | 4 (4) | 2 (3)
Dizziness (Nervous system disorders) | 18 (28) | 8 (12) | 2 (6)
Dysaesthesia (Nervous system disorders) | 1 (1) | 3 (7) | 0 (0)
Dysgeusia (Nervous system disorders) | 14 (32) | 3 (3) | 4 (6)
Headache (Nervous system disorders) | 8 (14) | 5 (6) | 4 (6)
Neurotoxicity (Nervous system disorders) | 3 (6) | 2 (2) | 2 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 17 (30) | 0 (0) | 3 (8)
Somnolence (Nervous system disorders) | 4 (8) | 1 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 5 (8) | 1 (1) | 1 (1)
Lacrimation increased (Eye disorders) | 4 (6) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 4 (8) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 5 (6) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (14) | 1 (1) | 8 (22)
Abdominal pain upper (Gastrointestinal disorders) | 10 (18) | 2 (3) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 4 (10) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 33 (80) | 10 (18) | 9 (17)
Diarrhoea (Gastrointestinal disorders) | 30 (66) | 3 (5) | 9 (28)
Dry mouth (Gastrointestinal disorders) | 14 (35) | 1 (2) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 8 (13) | 0 (0) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 5 (9) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 4 (5) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (17) | 1 (1) | 1 (2)
Haemorrhoids (Gastrointestinal disorders) | 4 (7) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 45 (158) | 19 (49) | 14 (64)
Vomiting (Gastrointestinal disorders) | 26 (79) | 12 (37) | 9 (21)
Alopecia (Skin and subcutaneous tissue disorders) | 38 (80) | 7 (8) | 10 (18)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (19) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 5 (8) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (8) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (9) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (19) | 2 (2) | 4 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (23) | 6 (11) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (8) | 2 (9) | 4 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (19) | 0 (0) | 3 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (11) | 1 (3) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 44 (143) | 16 (36) | 6 (14)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (13) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (9) | 2 (3) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 (14) | 0 (0) | 1 (35)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 2 (6) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 0 (0) | 1 (2)
Oral candidiasis (Infections and infestations) | 2 (3) | 1 (1) | 2 (4)
Paronychia (Infections and infestations) | 4 (6) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (3) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (9) | 1 (1) | 2 (3)
Urinary tract infection (Infections and infestations) | 7 (11) | 2 (3) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (3)
Proctalgia (Gastrointestinal disorders) | 1 (4) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (3)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (4) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (3) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebellar ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Intention tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (5)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0) | 2 (4)
Nail ridging (Skin and subcutaneous tissue disorders) | 3 (6) | 0 (0) | 1 (2)
Onycholysis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (2)
Palmar-plantar erythrodyaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 2 (3)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (2) | 0 (0) | 1 (3)
Hypertension (Vascular disorders) | 3 (5) | 1 (3) | 1 (2)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2014-10-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT01970540/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT01970540/SAP_001.pdf